CLINICAL TRIAL: NCT05389150
Title: Pharmacokinetic Non-interaction Study Between Pregabalin 150 Mg and Tramadol 50 Mg, Administered Individually or in Combination, Single Dose in Healthy Subjects of Both Genders Under Fasting Conditions
Brief Title: Non-interaction Study Between Pregabalin and Tramadol, Administered Individually or Combination, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BD PT-Sil No. 97-17
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Bioavailability; Fixed dose combination; Pregabalin; Tramadol; Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Tramadol; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Pregabalin/ Tramadol Fixed dose (Experimental): Pharmaceutical Form: Tablet Dosage: 150 mg / 50 mg Administration way: oral
  Interventions: Drug: Fixed dose combination Pregabalin 150 mg / Tramadol 50 mg
- Group B: Pregabalin (Lyrica®) (Active Comparator): Pharmaceutical Form: Capsule Dosage: 150 mg Administration way: oral
  Interventions: Drug: Pregabalin 150mg
- Group C: Tramadol (Tradol®) (Active Comparator): Pharmaceutical Form: Tablet Dosage: 50 mg Administration way: oral
  Interventions: Drug: Tramadol 50 mg

INTERVENTIONS:
Drug: Fixed dose combination Pregabalin 150 mg / Tramadol 50 mg — Pregabalin/Tramadol (Laboratorios Silanes S.A. de C.V.), Pharmaceutical Form: Tablet Dosage: 150 mg / 50 mg Administration way: oral
  Other Names: P/T
  Arms: Group A: Pregabalin/ Tramadol Fixed dose
Drug: Pregabalin 150mg — From Pfizer S.a. de C.V. Pharmaceutical Form: Capsule Dosage: 150 mg Administration way: oral
  Other Names: Preg (Lyrica®)
  Arms: Group B: Pregabalin (Lyrica®)
Drug: Tramadol 50 mg — From Grünenthal de México, S.A. de C.V. Pharmaceutical Form: Capsule Dosage: 50 mg Administration way: oral
  Other Names: Tram (Tradol®)
  Arms: Group C: Tramadol (Tradol®)

SUMMARY:
The study was carried out in the Clinical Unit and Analytical Unit of the Department of Pharmacology and Toxicology of the Faculty of Medicine of the Universidad Autónoma de Nuevo León, with the aim of comparing the bioavailability (maximum concentration and area under the curve) of an oral formulation containing Pregabalin 150 mg/Tramadol 50 mg in combination with the two oral formulations Pregabalin 150 mg or Tramadol 50 mg administered as a single dose, in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
The study design was crossover, 3 x 6 x 3, prospective and longitudinal, at a single dose of the combination Pregabalin 150 mg/Tramadol 50 mg administered orally versus each component administered individually, with three treatments, three periods, six sequences and one elimination period (wash out) of 7 days in 30 healthy subjects, under fasting conditions. The objective of the study was to characterize the pharmacokinetic parameters, maximum plasma concentration (Cmax), area under the curve (AUC), time to achieve Cmax (tmax), elimination constant (Ke), and elimination half life (t1/2) of Pregabalin and Tramadol after single oral dose administration, in combination: Pregabalin 150 mg/Tramadol 50 mg, tablets (Laboratorios Silanes S.A. de C.V.) versus each component individually managed, as well as to establish the frequency and type of events presented after the administration of a single dose of the formulations.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have been accepted by the COFEPRIS research subjects registration database.
* Subjects without a subordinate relationship with the researchers.
* Subjects who have given informed consent in writing.
* Subjects of both genders, aged between 18 and 55 years, Mexicans. - -Subjects with no background of hypersensitivity or allergies to the drug under study or related drugs.
* Body mass index between 18 and 27 kg/m2.
* Healthy subjects, according to the results of the complete clinical history, electrocardiogram and the integration of the results of the clinical analyses, carried out in certified clinical laboratories, without alterations that require a medical intervention as a consequence.
* Subjects with negative results for immunological tests (Anti-HIV, Anti-hepatitis B and C, VDRL).
* Subjects with negative results in drug abuse screening tests: tetrahydrocannabinoids, cocaine and amphetamines.
* Negative (qualitative) pregnancy test for women of childbearing potential without bilateral tubal obstruction or hysterectomy.
* In the case of women of childbearing age, they must have a birth control method, including barrier methods, non-hormonal intrauterine device, or bilateral tubal obstruction.

Exclusion Criteria:

* Subjects with recent history or physical examination evidence of gastrointestinal, renal, hepatic, endocrine, respiratory, cardiovascular, dermatological, or hematological disease that could affect the pharmacokinetic study of the product in research.
* Subjects who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken drugs potentially toxic within 30 days before the start of the study.
* Subjects who have received any medication during the 7 days before the start of the study.
* Subjects who have been hospitalized for any problem during the three months before the start of the study.
* Subjects who have been rejected by the registry database of research subjects of COFEPRIS, for having participated in a clinical study within the three months prior to the start of the study.
* Subjects who have received investigational drugs within the previous 60 days th the start of the study.
* Subjects allergic to the study drug or related drugs.
* Subjects who have ingested alcohol or drinks containing xanthines (coffee, tea, cocoa, chocolate, cola) or who have eaten charcoal-grilled food or grapefruit juice , at least 10 hours before the start of the study or who have smoked tobacco 24 hours before to the start of the internment period.
* Subjects who have donated or lost 450 mL or more of blood within the previous 60 days of the beginning of the study.
* Subjects with a history of drug and/or alcohol abuse according to the DSM-IV-TR Criteria.
* Research subjects who presents alterations in the vital signs recorded during the selection.
* Subjects who have consumed grapefruit or cranberry juice in the 10 hours prior to the study.
* Research subject with alterations of the vital signs recorded during the selection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose Pregabalin/Tramadol, employing the maximum observed concentration following the treatment (Cmax), obtained graphically, from the plasma concentration profile with respect to time.
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Pregabalin/Tramadol, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t) using the linear trapezoidal method.
The area under the curve from time zero to infinity calculated (AUC 0-inf) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Pregabalin/Tramadol, employing the area under the curve from time zero to infinity calculated (AUC 0-inf).
Time of the maximum measured concentration (Tmax) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Pregabalin/Tramadol, employing time of the maximum measured concentration (tmax), Obtained graphically, from the plasma concentration profile with respect to time.
Elimination rate (Ke) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Pregabalin/Tramadol, employing the elimination rate (Ke), estimated from the terminal linear portion of the plasma concentration profile with respect to time (on a semi-log scale)
Half time elimination (t1/2) | Baseline, 0.16, 0.33, 0.50, 1.00, 1.50, 2.0, 2.5, 3.0, 3.5, 4.0, 6.0, 10.0, 14.0, 24.0 and 36.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose Pregabalina/Tramadol, employing the half time elimination (t1/2) by the quotient of Ln(2)Ke.

SECONDARY OUTCOMES:
Frequency of occurrence of adverse events | 6 and 19 days
  The percentage of frequency of appearance of each adverse event was evaluated.
Adverse events | 6 and 19 days
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocaña, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel BN, Sharma N, Sanyal M, Shrivastav PS. An accurate, rapid and sensitive determination of tramadol and its active metabolite O-desmethyltramadol in human plasma by LC-MS/MS. J Pharm Biomed Anal. 2009 Feb 20;49(2):354-66. doi: 10.1016/j.jpba.2008.10.030. Epub 2008 Nov 5. PMID 19062215
- [Background] Filipe A, Almeida S, Pedroso PF, Neves R, Marques S, Sicard E, Massicotte J, Ortuno J. Single-Dose, Randomized, Open-Label, Two-Way, Crossover Bioequivalence Study of Two Formulations of Pregabalin 300 mg Hard Capsules in Healthy Volunteers Under Fasting Conditions. Drugs R D. 2015 Jun;15(2):195-201. doi: 10.1007/s40268-015-0094-8. PMID 25939332
- [Background] Zhou X, Liu J. Fluorescence detection of tramadol in healthy Chinese volunteers by high-performance liquid chromatography and bioequivalence assessment. Drug Des Devel Ther. 2015 Feb 26;9:1225-31. doi: 10.2147/DDDT.S73723. eCollection 2015. PMID 25750519
- [Background] Ben-Menachem E. Pregabalin pharmacology and its relevance to clinical practice. Epilepsia. 2004;45 Suppl 6:13-8. doi: 10.1111/j.0013-9580.2004.455003.x. PMID 15315511
- [Background] Zareba G. Pregabalin: a new agent for the treatment of neuropathic pain. Drugs Today (Barc). 2005 Aug;41(8):509-16. doi: 10.1358/dot.2005.41.8.910482. PMID 16234874
- [Background] Silva Mde F, Schramm SG, Kano EK, Mori Koono EE, Porta V, dos Reis Serra CH. Bioequivalence evaluation of single doses of two tramadol formulations: a randomized, open-label, two-period crossover study in healthy Brazilian volunteers. Clin Ther. 2010 Apr;32(4):758-65. doi: 10.1016/j.clinthera.2010.03.016. PMID 20435245
- [Background] Liu P, Liang S, Wang BJ, Guo RC. Development and validation of a sensitive LC-MS method for the determination of tramadol in human plasma and urine. Eur J Drug Metab Pharmacokinet. 2009 Jul-Sep;34(3-4):185-92. doi: 10.1007/BF03191172. PMID 20166437